CLINICAL TRIAL: NCT01719354
Title: Aftercare in the Community Health Center - a Venue for Identifying and Coordinating Community Services
Brief Title: Aftercare in the Community Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1770
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Mental Disorders
Keywords: Community Mental Health Centers; Norway; Aftercare
MeSH Terms: conditions — Mental Disorders | interventions — Community Health Centers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Health center (Experimental): Aftercare in a community Health center
  Interventions: Other: Community Health center
- Control (Active Comparator): AFtercare as usual in hospital/Mental health centers of District Psychiatric Service (DPS.
  Interventions: Other: Control

INTERVENTIONS:
Other: Community Health center — Observation of the functioning and coordination of health care before discharge to own home.
  Arms: Community Health center
Other: Control — standard aftercare in hospital/mental health centers of District Psychiatric Service (DPS).
  Arms: Control

SUMMARY:
This is a trial to examine the effects of aftercare for mental health patients in community health center (Leistad). Recruitment occurs among hospitalized patients in psychiatric hospitals (Østmarka). After discharge, patients will be randomly assigned to one of two groups: intervention group (community health center, primary care) or control group (Community mental health centers of District Psychiatric Service, specialist care).

The project's primary objective is to investigate the effect of community services on patients' functional capacity and user satisfaction after discharge. Secondly, the number of treatment days and readmissions to mental health care will be examined. The project will also compare costs of hospitalization, in psychiatric hospital and community health center respectively. Data will be collected from community health records, medical records and patient systems in psychiatric hospital, community mental health centers of District Psychiatric Service (DPS) and questionnaires filled out by patients.

ELIGIBILITY:
Inclusion Criteria:

* considered by the responsible manager to have given consent
* hospitalized, diagnosed and treated such as can be continued in a District Psychiatric Service or a health center.
* stable condition, but anxiety and disruptive behavior may occur to a lesser extent.
* considered to have a perceived need for complex services from specialist health and community for a long time after discharge.

Exclusion Criteria:

* not in a stable phase thus shielding required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Consumption of community health service | one year
  Measure different types of community health services in hours per week.
Need for community health services | one year
  Using IPLOS (Norw. individual-based nursing and care statistics) form with 17 variables to identify patient needs
User satisfaction | one year
  A qualitative analysis of interviews of 10 patients who have been admitted to the District Psychiatric Service and community health center.
Need for community health services | one year
  Using individual-based nursing and care statistics (Norw. IPLOS) form with 17 variables to identify patient needs

SECONDARY OUTCOMES:
Number of treatment days | One year
  Number of treatment days in hospital and District Psychiatric Service compared with number of treatment days in community health center.
Readmission | One year
  Readmission in hospital.
The total costs of inpatient and total costs of all health care after discharge | One year
  Costs per day in hospital; Costs per day for District Psychiatric Service; Costs per day in community health center

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, prof, Study Director — NTNU, Department of Public Health and General Practice
Locations (1):
- Regional Committees for Medical and Health Research Ethics, Trondheim, Norway

REFERENCES:
- [Derived] Roos E, Bjerkeset O, Steinsbekk A. Health care utilization and cost after discharge from a mental health hospital; an RCT comparing community residential aftercare and treatment as usual. BMC Psychiatry. 2018 Nov 12;18(1):363. doi: 10.1186/s12888-018-1941-2. PMID 30419894